CLINICAL TRIAL: NCT02477527
Title: Switching From Atripla to Stribild Leads to Improvements in Central Nervous System Side Effects and Sleep Disturbances
Brief Title: Atripla to Stribild Switch Study to Evaluate Sleep Disturbances
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Midtown Medical Center, Tampa, FL (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB001JP001
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: HIV; AIDS; Sleep Disorders
Keywords: atripla; stribild; dreams
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sleep Wake Disorders | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stribild (Experimental): Patients to be changed from Atripla to elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil and observed for changes in sleep patterns / sleep disturbances.
  Interventions: Drug: Stribild

INTERVENTIONS:
Drug: Stribild — Change subjects from Atripla one tablet per day to elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil one tablet per day.

SUMMARY:
Switch patients from Atripla to Stribild will be evaluated to see if patients have less sleep disturbances.

DETAILED DESCRIPTION:
Stribild is a preferred regimen in the Department of Health and Human Services guidelines and has demonstrated non-inferiority to Atripla in treatment naïve patients out to 144 weeks (GS-102). Stribild also has statistically significant less Central Nervous System side effects, sleep disturbances and lipid elevations compared to Atripla. This study will evaluate the efficacy, safety, changes in Central Nervous System abnormalities and sleep disorders following a switch from virologically suppressed subjects on Atripla to Stribild.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ subjects 18 years of age or older
* estimated Glomerular Filtration Rate > 70 mL/min
* must currently be on Atripla and taking it for at least 3 months with a HIV-1 Viral Load < 50 copies/mL
* no antiretrovirals prior to the initiation of Atripla
* baseline genotyping

Exclusion Criteria:

* pregnancy
* unable to provide informed consent
* enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Braun, MD, Principal Investigator — Midtown Medical Center

IPD SHARING:
Plan to Share IPD: No
can be obtained by contacting the investigator only.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from private office practice.
Pre-assignment Details: Participants had to be stable on Atripla for at least 6 months with undetectable viral load.
Groups:
- Study: Patients to be changed from Atripla to elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil and observed for changes in sleep patterns / sleep disturbances.
  elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil: Change subjects from Atripla one tablet per day to elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil one tablet per day.
Period: Overall Study
Arm/Group | Study
Started | 27
Completed | 21
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 3

BASELINE CHARACTERISTICS:
Groups:
- Stribild: Patients to be changed from Atripla to elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil and observed for changes in sleep patterns / sleep disturbances.
  elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil: Change subjects from Atripla one tablet per day to elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil one tablet per day.
Arm/Group | Stribild
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participants in years at time of enrollment
  years | 48.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Private practice office located in Tampa, Florida.
  participants
    United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Viral Loads < 50 Following the Switch
Description: percentage of patients with viral loads < 50 following the switch at 24 weeks.
Time Frame: 24 weeks
Population: Participants completing the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Study
Number analyzed (Participants) | 21
Participants | 20

2. Secondary Outcome: T-cell Changes
Description: Change in CD4 Cell count from baseline to 24 weeks.
Time Frame: 24 weeks
Population: Participants completing the study.
Measure: Mean (Full Range); unit: cells / cc
Arm/Group | Study
Number analyzed (Participants) | 21
cells / cc | 151 [5 to 644]

3. Secondary Outcome: Improvements in Central Nervous System Toxicity Score
Description: Changes in Central Nervous System toxicity score at week 24 as measured by SSAT 047 scale.
  The scale is a questionnaire that participants complete at each visit. The SSAT 047 scores 10 items related to efavirenz side effects including: dizziness, depression, insomnia, anxiety, confusion, impaired concentration, headache, somnolence, aggressive mood and abnormal dreams. The side effects were scored as 0 for "None", 1 for "Mild", 2 for "Moderate" and 3 for "Severe". The scores for the 10 items ranged from 0(none) - 3(severe), and the total score is 0-30. The scores are then averaged to determine the overall impact on central nervous system symptoms and reported as the sum of the measures.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Study
Number analyzed (Participants) | 21
units on a scale | 2.0 [-1.0 to 3.0]

4. Secondary Outcome: Improvements in Sleep Disorder Score
Description: Changes in quality of sleep at week 24 as measured by Pittsburgh Sleep Quality Index (PSQI). The Pittsburgh Sleep Quality Index (PSQI) is used to measure the quality and patterns of sleep in adults. It rates sleep based on seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. It is a self-administered questionnaire covering these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. The scores for the 7 items ranged from 0(none) - 3(severe), and the total score is 0-21. The reported values in the table represent the change in the overall scores on the PSQI scale. The values were added and reported as the sum of the individual measures. A negative score correlates with improvement of the sleep quality.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Study
Number analyzed (Participants) | 21
units on a scale | -4 [-17 to 3]

5. Other Pre Specified Outcome: Safety as Measured by Side Effects
Description: Monitor for any side effects that are spontaneously reported by subjects and reported on questionnaires.
Time Frame: 24 weeks
Population: no adverse effects reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Study
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 month duration of the study
Description: Adverse events were solicited from patients.
Arm/Group | Study
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No